CLINICAL TRIAL: NCT03054298
Title: Phase I Study of Human Chimeric Antigen Receptor Modified T Cells in Patients With Mesothelin Expressing Cancers
Brief Title: CAR T Cells in Mesothelin Expressing Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Tmunity Therapeutics, a wholly owned subsidiary of Kite Pharma (a Gilead company) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 826085 (UPCC 02916)
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Lung Adenocarcinoma; Ovarian Cancer; Peritoneal Carcinoma; Fallopian Tube Cancer; Mesotheliomas Pleural; Mesothelioma Peritoneum
MeSH Terms: conditions — Adenocarcinoma of Lung; Ovarian Neoplasms; Fallopian Tube Neoplasms; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Active Comparator): Single dose of 1-3x10^7 huCARTmeso cells/m^2
  Interventions: Biological: huCART-meso cells
- Cohort 2 (Active Comparator): Cyclophosphamide 1 gram/m^2 administered 2-4 days prior to a single dose of 1-3x10^7 huCARTmeso cells/m^2
  Interventions: Biological: huCART-meso cells
- Cohort 3 (Active Comparator): PERMANENTLY CLOSED
  Interventions: Biological: huCART-meso cells
- Cohort 4 (Active Comparator): PERMANENTLY CLOSED
  Interventions: Biological: huCART-meso cells
- Cohort 5 (Active Comparator): Single dose of 1-3x10^7 huCART-meso cells/m^2 day 0 by intrapleural infusion (IP) through an indwelling pleural catheter without any conditioning chemotherapeutic regimen.
  Interventions: Biological: huCART-meso cells
- Cohort 6 (Active Comparator): Cyclophosphamide 1 gram/m^2 administered 2-4 days prior to dose of 1-3x10^7 huCART-meso cells/m^2 via IV infusion on Day 0. This initial infusion may be followed by up to two additional IV infusions of huCART-meso cells at the same dose level, given approximately 21-42 days apart, if the subject meets eligibility to receive additional infusions. Cyclophosphamide will not be repeated prior to subsequent doses of huCART-meso cells.
  Interventions: Biological: huCART-meso cells
- Cohort 7 (Active Comparator): Cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day given over 3 days by IV infusion followed by a single dose of 1-3x10^7 huCART-meso cells/m^2 via intraperitoneal (i.p.) administration. Lymphodepleting chemotherapy will be scheduled such that the last day of chemotherapy is 3 days (+/- 1 day) prior to the infusion of huCART-meso cells. This initial i.p. infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart. The subject must meet eligibility to receive additional infusions. Lymphodepleting chemotherapy will not be repeated prior to additional infusions of huCART-meso cells.
  Interventions: Biological: huCART-meso cells

INTERVENTIONS:
Biological: huCART-meso cells — Intravenous administration or local delivery of lentiviral transduced huCART-meso cells in 7 cohorts with or without lymphodepletion..

SUMMARY:
Phase I study to establish safety and feasibility of both intravenous administration and local delivery of lentiviral transduced huCART-meso cells with or without lymphodepletion.

DETAILED DESCRIPTION:
This is a Phase I study evaluating the safety and feasibility of both intravenous administration and local delivery of lentiviral transduced huCART-meso cells with and without lymphodepleting chemotherapy.

* Cohort 1 (N=3-6): will receive a single dose of 1-3x10^7 huCARTmeso cells/m^2 on day 0 without any conditioning chemotherapeutic regimen.
* Cohort 2 (N=3-6): will receive a single dose of 1-3x10^7 huCARTmeso cells/m^2 on day 0, following a flat dose of 1 gram/m2 of cyclophosphamide administered 2-4 days prior to huCARTmeso cells (day -4 to day -2).
* Cohort 3 (N=3-6): will receive a single dose of 1-3x10^8 /m^2 lentiviral transduced huCART-meso cells on day 0 without any conditioning chemotherapeutic regimen. **Cohort 3 permanently closed**
* Cohort 4 subjects (N=3-6) will receive a single dose of 1-3x10^8 /m^2 lentiviral transduced huCART-meso cells on day 0, following a flat dose of 1 gram/m^2 of cyclophosphamide administered 2-4 days prior to huCART-meso cells (day -4 to day -2). **Cohort 4 permanently closed**
* Cohort 5 (N=up to 6): will receive a single dose of 1-3x10^7 huCARTmeso cells/m^2 on day 0 by intrapleural infusion (IP) through an indwelling pleural catheter without any conditioning chemotherapeutic regimen. The safety of this dose level has been established by Cohorts 1 and 2.
* Cohort 6 (N=up to 6): will receive a dose of 1-3x10^7 huCARTmeso cells/m^2 via IV infusion on Day 0, following a flat dose of 1 gram/m^2 of cyclophosphamide administered 2-4 days prior to huCART-meso cells (~Day -4 to -2). This initial infusion may be followed by up to two additional IV infusions of huCART-meso cells at the same dose level, given between 21-42 days apart, if the subject meets eligibility to receive additional infusions. Cyclophosphamide will not be repeated prior to subsequent doses of huCART-meso cells. Enrollment into Cohort 6 will occur in parallel with Cohort 5.
* Cohort 7 (N = up to 6): will receive a single dose of 1-3x10^7 huCART-meso cells/m^2 via intraperitoneal (i.p.) administration, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m^2/day and fludarabine 30 mg/m^2/day given over 3 days by intravenous infusion. Lymphodepleting chemotherapy will be scheduled such that the last day of chemotherapy is 3 days (+/- 1 day) prior to the 1st infusion of huCART-meso cells. This initial i.p. infusion may be followed by up to two additional infusions of huCART-meso cells via intravenous (IV) administration at the same dose level, given between 21-42 days apart. The subject must meet eligibility to receive additional infusions. Lymphodepleting chemotherapy will not be repeated prior to additional infusions of huCART-meso cells.

The Maximum Tolerated Dose (MTD) is defined as the dose at which 0-1 DLT occurs in 6 evaluable subjects tested within the dose range of this study. The maximum tolerated dose has been established as 1-3x10^7 huCARTmeso cells/m^2.

Adverse events will be collected and evaluated during the protocol specified adverse event reporting period

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed cancer (one of the following):

   1. Cohorts 1-4 and Cohort 6 participants:

      **Note: Cohorts 3 and 4 permanently closed**
      * Metastatic or recurrent lung adenocarcinoma.
      * Persistent or recurrent serous epithelial ovarian cancer or primary peritoneal carcinoma or fallopian tube carcinoma
      * Malignant pleural and peritoneal mesothelioma (histologically confirmed epithelial)
   2. Cohort 5 participants: **Note: As of 1-Feb-2021 lung adenocarcinoma patients are no longer being enrolled in this trial**

      * Metastatic or recurrent lung adenocarcinoma with documented pleural effusion
      * Persistent or recurrent serous epithelial ovarian cancer or primary peritoneal carcinoma or fallopian tube carcinoma with documented pleural effusion
      * Malignant pleural and peritoneal mesothelioma (histologically confirmed epithelial) with documented pleural effusion
   3. Cohort 7 patients:

      * Persistent or recurrent serous epithelial ovarian cancer or primary peritoneal carcinoma or fallopian tube carcinoma with evidence of ascites
      * Malignant peritoneal mesothelioma (histologically confirmed epithelial)
2. CRITERIA HAS BEEN RETIRED
3. Failure of at least one prior standard of care chemotherapy for advanced stage disease. ALLOWANCE FOR PRIOR PD-1 or PDL-1 THERAPIES REMOVED.
4. Patients must have measurable disease as defined by RECIST 1.1 criteria or modified RECIST criteria (mesothelioma only).
5. Subjects with asymptomatic CNS metastases that have been treated (and are off steroids for the treatment of CNS disease) are allowed. They must meet the following at the time of enrollment:

   1. No concurrent treatment for the CNS disease
   2. No progression of CNS metastasis on MRI at screening scans
   3. No evidence of leptomeningeal disease or cord compression
6. Subjects ≥ 18 years of age.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Satisfactory organ and bone marrow function as defined by the following:

   * Absolute neutrophil count ≥ 1,000/μl
   * Platelets ≥75,000/μl
   * Hemoglobin ≥ 8 g/dL
   * Direct bilirubin ≤ 2.0 mg/dl unless secondary to bile duct obstruction by tumor or Gilbert's syndrome with a direct bilirubin of less that 3.0 mg/dl is allowed.
   * Creatinine ≤ 1.5x the institutional normal upper limit
   * Albumin ≥ 2
   * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 5x the institutional normal upper limit
   * Cardiac ejection fraction of ≥40% as measured by resting echocardiogram, with no clinically significant pericardial effusion.
9. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT ≤ 1.2 time the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
10. Provide written informed consent.
11. Subjects of reproductive potential must agree to use acceptable birth control methods.

Exclusion Criteria

1. Sarcomatoid and biphasic mesothelioma.
2. Known leptomeningeal carcinomatosis or spinal cord compression. Screening for this is not required unless suspicious symptoms.
3. Subjects with symptomatic CNS metastases are excluded.
4. EXCLUSION CRITERIA HAS BEEN RETIRED
5. Active invasive cancer other than the one of the three cancers in this study. Subjects with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder and prostate cancer with PSA level < 1.0) are not excluded.
6. HIV infection
7. Active hepatitis B or hepatitis C infection
8. Active autoimmune disease (including but not limited to: systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within four (4) weeks prior to eligibility confirmation by physician-investigator, with the exception of thyroid replacement.
9. Patients with ongoing or active infection.
10. Dependence on systemic steroids or immunosupressant medications.
11. Patients requiring supplemental oxygen therapy.
12. Prior therapy with lentiviral gene modified cells.
13. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
14. Any clinically significant pericardial effusion, Class II-IV cardiovascular disability according to the New York Heart Association Classification or other cardiovascular condition that would preclude assessment of mesothelin induced pericarditis, or which may worsen as a result of expected toxicities in this study. This determination will be made by a cardiologist if cardiac issues are suspected.
15. Any clinically significant pleural or peritoneal effusion that cannot be drained with standard approaches. An indwelling drainage device placed prior to eligibility confirmation by physician / investigator is acceptable.
16. Pregnant or breastfeeding women.
17. EXCLUSION HAS BEEN RETIRED
18. EXCLUSION HAS BEEN RETIRED
19. Subjects with significant lung disease as follows:

    * Subjects with radiographic evidence of greater than lobar lymphangitic pulmonary involvement, greater than lobar bronchial wall thickening suggestive of peribronchial lymphatic disease extension, and/or evidence of extensive bilateral parenchymal metastatic burden.
    * Subjects with radiographic and/or clinical evidence of active radiation pneumonitis.
    * Subjects with radiographic evidence of underlying interstitial lung disease, including evidence of unresolved drug toxicity from any agent (e.g. chemotherapy, targeted agents, amiodarone, nitrofurantoin, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janos L Tanyi, MD, PhD, Principal Investigator — University of Pennaylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol specifies that a consented participant is an enrolled participant. 65 participants were consented. Of these, 34 were ineligible and 31 were eligible. Of the 31 eligible, one participant was never assigned to a cohort. This participant was withdrawn prior to assignment due to disease progression.
  The remaining 30 participants are detailed below.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Started | 3 | 3 | 2 | 0 | 6 | 8 | 8
Completed | 3 | 3 | 2 | 0 | 2 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Cohort 4 was permanently closed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7 | Total
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 6 | 8 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 |  | 6 | 6 | 6 | 24
  >=65 years | 0 | 1 | 1 |  | 0 | 2 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [54.5 to 63.2] | 62.3 [52.7 to 76.1] | 68.1 [61.9 to 74.3] |  | 61.1 [54.6 to 68.1] | 59.7 [39.1 to 72.8] | 63.0 [42.3 to 80.4] | 61.6 [39.1 to 80.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 |  | 5 | 7 | 8 | 27
  Male | 1 | 0 | 0 |  | 1 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 |  | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 2 | 2 |  | 6 | 8 | 8 | 29
  Unknown or Not Reported | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 |  | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 |  | 0 | 0 | 1 | 1
  White | 2 | 2 | 2 |  | 6 | 8 | 6 | 26
  More than one race | 0 | 0 | 0 |  | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 |  | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 2 |  | 6 | 8 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Time Frame: 7 years
Population: Cohort 4 closed prematurely.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 2 | 6 | 6
Participants | 3 | 3 | 2 | 0 | 2 | 6 | 6

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using RECIST V1.1 - at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression.
Time Frame: 7 years
Population: Cohort 4 was permanently closed.
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 2 | 6 | 6
weeks | 8.1 [4.1 to 13.1] | 7 [4 to 26] | 7.6 [0.7 to 14.4] |  | 13.5 [11 to 16] | 14.1 [8.4 to 96] | 12.3 [4 to 22.3]

3. Secondary Outcome: Overall Survival
Time Frame: 7 years
Population: Cohort 4 was prematurely closed.
Measure: Median (Full Range); unit: weeks
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 2 | 6 | 6
weeks | 14.6 [8.2 to 58.9] | 129.6 [9.7 to 145.7] | 57.9 [0.7 to 115] |  | 65.2 [49.3 to 81.1] | 81.1 [9.4 to 118] | 22 [18.3 to 32.4]

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate is the proportion of subjects in the efficacy-evaluable set with radiologically confirmed measurable disease at baseline, who achieved partial response (PR) or better after infusion as determined by RECIST 1.1. Missing or non-evaluable time points will not be included.
  Per RECIST 1.1, a complete response is defined as "disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm." A partial response is defined as "at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters."
Time Frame: Month 6
Population: Cohort 4 was permanently closed.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
Number analyzed (Participants) | 3 | 3 | 2 | 0 | 2 | 6 | 6
percentage of participants | 0 | 0 | 0 |  | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 7 years
Description: Cohort 4 was closed without any subjects being enrolled.
  Subjects were transitioned to a separate long-term follow-up (LTFU) protocol for a variety of reasons (e.g. disease progression, receipt of alternative therapy, PI discretion, etc). Only protocol-defined adverse events (PDAEs) were collected/reported on the separate LTFU protocol, and death due to disease progression was not considered a PDAE. PDAEs are defined in the protocol section 8.1.1.
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 6 | Cohort 7
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 0/0 | 2/2 | 4/6 | 6/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/2 | 0/0 | 1/2 | 4/6 | 6/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 2/2 | 0/0 | 2/2 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=2) | Cohort 4 (N=0) | Cohort 5 (N=2) | Cohort 6 (N=6) | Cohort 7 (N=6)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | NA | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | NA | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Other (Viral gastroenteritis) (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Edema limbs (General disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | NA | 0 | 1 | 0
Other (disease progression) (General disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Infusion related reaction (General disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Cytokine release syndrome (Infections and infestations) | 0 | 0 | 1 | NA | 1 | 2 | 4
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | NA | 0 | 1 | 0
Other (COVID-19) (Infections and infestations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | NA | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | NA | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Other (CAR Neurotoxicity) (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 0 | 2
Other (possible drug withdrawal) (Nervous system disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 1 | NA | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | NA | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 0 | 1 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2 | NA | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=2) | Cohort 4 (N=0) | Cohort 5 (N=2) | Cohort 6 (N=6) | Cohort 7 (N=6)
Anemia (Blood and lymphatic system disorders) | 2 | 2 | 1 | NA | 1 | 3 | 6
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | NA | 0 | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | NA | 1 | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Other (anisocoria) (Eye disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Other (burning sensation) (Eye disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | NA | 1 | 0 | 4
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Bloating (Gastrointestinal disorders) | 1 | 0 | 1 | NA | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 1 | NA | 0 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | NA | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | NA | 0 | 1 | 0
Other (Pain RUQ) (Gastrointestinal disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | NA | 1 | 5 | 5
Stomach pain (Gastrointestinal disorders) | 2 | 0 | 0 | NA | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | NA | 1 | 4 | 4
Chills (General disorders) | 1 | 0 | 0 | NA | 0 | 1 | 0
Edema limbs (General disorders) | 2 | 1 | 0 | NA | 0 | 1 | 2
Fatigue (General disorders) | 2 | 2 | 1 | NA | 1 | 3 | 4
Fever (General disorders) | 1 | 0 | 0 | NA | 0 | 0 | 2
Malaise (General disorders) | 1 | 1 | 0 | NA | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2 | 0 | NA | 1 | 3 | 0
Pain (General disorders) | 1 | 0 | 0 | NA | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Anaphylaxis (Immune system disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | NA | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | NA | 0 | 1 | 4
Other (Drug overdose) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | NA | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Alanine animotransferase increased (Investigations) | 0 | 0 | 0 | NA | 0 | 1 | 2
Alkaline phosphatase increased (Investigations) | 1 | 2 | 0 | NA | 0 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | NA | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
Creatinine increased (Investigations) | 1 | 0 | 1 | NA | 0 | 3 | 0
Fibrinogen decreased (Investigations) | 0 | 0 | 0 | NA | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 0 | NA | 0 | 1 | 2
Lymphocyte count decreased (Investigations) | 2 | 3 | 1 | NA | 1 | 6 | 6
Neutrophil count decreased (Investigations) | 0 | 2 | 0 | NA | 1 | 3 | 4
Platelet count decreased (Investigations) | 1 | 1 | 1 | NA | 0 | 1 | 4
Weight loss (Investigations) | 0 | 1 | 0 | NA | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 3 | 1 | NA | 1 | 5 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA | 0 | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | NA | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | NA | 0 | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | NA | 1 | 5 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | NA | 1 | 3 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | NA | 0 | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | 0 | 4 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 1 | NA | 0 | 3 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | NA | 0 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | NA | 1 | 2 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA | 0 | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 0 | 2 | 1
Ataxia (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 4 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0 | NA | 0 | 4 | 2
Paresthesia (Nervous system disorders) | 2 | 1 | 0 | NA | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | NA | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | NA | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | NA | 0 | 0 | 2
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | NA | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 1 | 0 | NA | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | NA | 1 | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | NA | 0 | 2 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 2 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | 1 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | NA | 0 | 1 | 0
Other (goose bumpy feeling) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | NA | 0 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 1 | 0 | NA | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | NA | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | NA | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03054298/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03054298/ICF_001.pdf